CLINICAL TRIAL: NCT00452153
Title: Evaluation of Legionella PCR Techniques for the Routine Diagnosis of Legionellosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Too much difficulties to includ patient
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0601072
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Legionellosis
Keywords: legionellosis; diagnosis of legionellosis; PCR
MeSH Terms: conditions — Legionellosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Characterization Legionnella (Experimental): Characterization Legionnella by polymerase chain reaction (PCR)
  Interventions: Procedure: Characterization Legionnella

INTERVENTIONS:
Procedure: Characterization Legionnella — * Characterisation Legionnella by polymerase chain reaction (PCR)
  * Characterization strain of Legionnella by sequencing the 23S-5S ribosomal intergenic spacer region

SUMMARY:
The validity of molecular techniques for the diagnosis of legionellosis is not known. Although PCR can detect Legionella pneumophila (responsible for 80% of legionellosis) and other Legionella species, this test is not recommended in standard guidelines to assess this diagnostic, by contrast to culture of sputum, serology and urine antigen. The aim of this study is to evaluate Legionella PCR techniques, performed directly onto the sputum aspirates, for the routine diagnosis of pneumonia in adults' patients admitted to hospital. This study implicates 3 University hospitals (Lyon, Grenoble and Saint-Etienne) in collaboration with the French reference center of legionellosis for a previous duration of one year. In addition to the usual diagnostic tests that are performed when pneumonia is suspected, real-time PCR will be added for the detection and differentiation of Legionella. Hypothesizing the inclusion of 1000 pneumonia in this study, the predictable number of newly-detected legionellosis will be approximately 60 to 70 cases. According to a predefined algorithm, cases of legionellosis will be classified as definite or probable. Sensitivity and specificity of the real-time PCR will be calculated according to this classification. This study is intended to validate real-time PCR as a tool for the rapid diagnosis of legionellosis, allowing to optimize the antibiotic treatment of pneumonia. PCR techniques can also contribute to the better detection and differentiation of Legionella sp infections that are not documented accurately by routine microbiologic tests.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patient affiliated to social insurance
* Community acquired or nosocomial pneumonia

Exclusion Criteria:

* No sputum aspirate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Definite or probable legionellosis | Inclusion and J30

SECONDARY OUTCOMES:
Definite legionellosis | Inclusion and J30
Probable legionellosis | Inclusion and J30
Possible legionellosis | Inclusion and J30

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Berthelot, PU-PH, Principal Investigator — CHU SAINT-ETIENNE
Locations (6):
- France (6):
  - HMU CHU Saint-Etienne, Saint-Etienne
  - Infectious Disease unit CHU de Saint-Etienne, Saint-Etienne
  - Pneumology unit CHU de Saint-Etienne, Saint-Etienne
  - Reanimation unit - Hopital Bellevue - CHU de Saint-Etienne, Saint-Etienne
  - Reanimation unit - Hôpital NORD - CHU de Saint-Etienne, Saint-Etienne
  - Urgency unit CHU Saint-Etienne, Saint-Etienne

REFERENCES:
- [Background] Squier CL, Stout JE, Krsytofiak S, McMahon J, Wagener MM, Dixon B, Yu VL. A proactive approach to prevention of health care-acquired Legionnaires' disease: the Allegheny County (Pittsburgh) experience. Am J Infect Control. 2005 Aug;33(6):360-7. doi: 10.1016/j.ajic.2005.01.012. PMID 16061143
- [Background] Decludt B, Campese C, Lacoste M, Che D, Jarraud S, Etienne J. Clusters of travel associated legionnaires' disease in France, September 2001- August 2003. Euro Surveill. 2004 Feb;9(2):12-3. doi: 10.2807/esm.09.02.00446-en. PMID 15010573
- [Background] Grattard F, Berthelot P, Reyrolle M, Ros A, Etienne J, Pozzetto B. Molecular typing of nosocomial strains of Legionella pneumophila by arbitrarily primed PCR. J Clin Microbiol. 1996 Jun;34(6):1595-8. doi: 10.1128/jcm.34.6.1595-1598.1996. PMID 8735131
- [Background] Aurell H, Etienne J, Forey F, Reyrolle M, Girardo P, Farge P, Decludt B, Campese C, Vandenesch F, Jarraud S. Legionella pneumophila serogroup 1 strain Paris: endemic distribution throughout France. J Clin Microbiol. 2003 Jul;41(7):3320-2. doi: 10.1128/JCM.41.7.3320-3322.2003. PMID 12843082
- [Background] Gaia V, Fry NK, Afshar B, Luck PC, Meugnier H, Etienne J, Peduzzi R, Harrison TG. Consensus sequence-based scheme for epidemiological typing of clinical and environmental isolates of Legionella pneumophila. J Clin Microbiol. 2005 May;43(5):2047-52. doi: 10.1128/JCM.43.5.2047-2052.2005. PMID 15872220
- [Background] Wang EE, Manson B, Corey M, Bernard K, Prober CG. False positivity of Legionella serology in patients with cystic fibrosis. Pediatr Infect Dis J. 1987 Mar;6(3):256-9. doi: 10.1097/00006454-198703000-00009. PMID 3106925
- [Background] Plouffe JF, File TM Jr, Breiman RF, Hackman BA, Salstrom SJ, Marston BJ, Fields BS. Reevaluation of the definition of Legionnaires' disease: use of the urinary antigen assay. Community Based Pneumonia Incidence Study Group. Clin Infect Dis. 1995 May;20(5):1286-91. doi: 10.1093/clinids/20.5.1286. PMID 7620012
- [Background] Helbig JH, Uldum SA, Bernander S, Luck PC, Wewalka G, Abraham B, Gaia V, Harrison TG. Clinical utility of urinary antigen detection for diagnosis of community-acquired, travel-associated, and nosocomial legionnaires' disease. J Clin Microbiol. 2003 Feb;41(2):838-40. doi: 10.1128/JCM.41.2.838-840.2003. PMID 12574296
- [Background] Grattard F, Ginevra C, Riffard S, Ros A, Jarraud S, Etienne J, Pozzetto B. Analysis of the genetic diversity of Legionella by sequencing the 23S-5S ribosomal intergenic spacer region: from phylogeny to direct identification of isolates at the species level from clinical specimens. Microbes Infect. 2006 Jan;8(1):73-83. doi: 10.1016/j.micinf.2005.05.022. Epub 2005 Aug 8. PMID 16198139
- [Background] Hayden RT, Uhl JR, Qian X, Hopkins MK, Aubry MC, Limper AH, Lloyd RV, Cockerill FR. Direct detection of Legionella species from bronchoalveolar lavage and open lung biopsy specimens: comparison of LightCycler PCR, in situ hybridization, direct fluorescence antigen detection, and culture. J Clin Microbiol. 2001 Jul;39(7):2618-26. doi: 10.1128/JCM.39.7.2618-2626.2001. PMID 11427579
- [Background] Templeton KE, Scheltinga SA, Sillekens P, Crielaard JW, van Dam AP, Goossens H, Claas EC. Development and clinical evaluation of an internally controlled, single-tube multiplex real-time PCR assay for detection of Legionella pneumophila and other Legionella species. J Clin Microbiol. 2003 Sep;41(9):4016-21. doi: 10.1128/JCM.41.9.4016-4021.2003. PMID 12958219
- [Background] Welti M, Jaton K, Altwegg M, Sahli R, Wenger A, Bille J. Development of a multiplex real-time quantitative PCR assay to detect Chlamydia pneumoniae, Legionella pneumophila and Mycoplasma pneumoniae in respiratory tract secretions. Diagn Microbiol Infect Dis. 2003 Feb;45(2):85-95. doi: 10.1016/s0732-8893(02)00484-4. PMID 12614979
- [Background] Reischl U, Linde HJ, Lehn N, Landt O, Barratt K, Wellinghausen N. Direct detection and differentiation of Legionella spp. and Legionella pneumophila in clinical specimens by dual-color real-time PCR and melting curve analysis. J Clin Microbiol. 2002 Oct;40(10):3814-7. doi: 10.1128/JCM.40.10.3814-3817.2002. PMID 12354888
- [Background] Ginevra C, Barranger C, Ros A, Mory O, Stephan JL, Freymuth F, Joannes M, Pozzetto B, Grattard F. Development and evaluation of Chlamylege, a new commercial test allowing simultaneous detection and identification of Legionella, Chlamydophila pneumoniae, and Mycoplasma pneumoniae in clinical respiratory specimens by multiplex PCR. J Clin Microbiol. 2005 Jul;43(7):3247-54. doi: 10.1128/JCM.43.7.3247-3254.2005. PMID 16000443
- [Background] Helbig JH, Bernander S, Castellani Pastoris M, Etienne J, Gaia V, Lauwers S, Lindsay D, Luck PC, Marques T, Mentula S, Peeters MF, Pelaz C, Struelens M, Uldum SA, Wewalka G, Harrison TG. Pan-European study on culture-proven Legionnaires' disease: distribution of Legionella pneumophila serogroups and monoclonal subgroups. Eur J Clin Microbiol Infect Dis. 2002 Oct;21(10):710-6. doi: 10.1007/s10096-002-0820-3. Epub 2002 Oct 18. PMID 12415469
- [Background] Wellinghausen N, Frost C, Marre R. Detection of legionellae in hospital water samples by quantitative real-time LightCycler PCR. Appl Environ Microbiol. 2001 Sep;67(9):3985-93. doi: 10.1128/AEM.67.9.3985-3993.2001. PMID 11525995
- [Background] Woodhead M. Community-acquired pneumonia in Europe: causative pathogens and resistance patterns. Eur Respir J Suppl. 2002 Jul;36:20s-27s. doi: 10.1183/09031936.02.00702002. PMID 12168744